CLINICAL TRIAL: NCT04490993
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Phase Ⅲ Clinical Trial to Evaluate the Clinical Safety and Efficacy of APL-1202 in Combination With Epirubicin Hydrochloride Versus Epirubicin Hydrochloride Alone in Intermediate and High-risk Chemo-refractory Non-muscle Invasive Bladder Cancer (NMIBC) Patients
Brief Title: Safety and Efficacy of APL-1202 in Combination With Epirubicin Hydrochloride Versus Epirubicin Hydrochloride Alone in Intermediate and High-risk Chemo-refractory Non-muscle Invasive Bladder Cancer (NMIBC) Patients
Acronym: ACCRUE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu Yahong Meditech Co., Ltd aka Asieris (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YHCT-NIT-R1
Record Dates: First submitted 2020-07-23; First posted 2020-07-29 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Non-muscle Invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Epirubicin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- APL-1202 treatment (Experimental)
  Interventions: Drug: APL-1202 in combination with Epirubicin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo in combination with Epirubicin

INTERVENTIONS:
Drug: APL-1202 in combination with Epirubicin — * Induction period: APL-1202 is administered for 12 consecutive weeks
  * Maintenance period: after 12-week drug free period, APL-1202 is administered for another12 consecutive weeks as maintenance treatment
  * Follow up period: APL-1202 is administered at every 3-month interval if no events occurred in the treatment period and until the occurrence of events or the end of the entire clinical trial Intravesical Epirubicin hydrochloride will be administered once weekly for consecutive 6-8 weeks in the induction period, followed by once monthly in the maintenance period until end of 12 months
  Arms: APL-1202 treatment
Drug: Placebo in combination with Epirubicin — * Induction period: placebo is administered for 12 consecutive weeks
  * Maintenance period: after 12-week drug free period, placebo is administered for another12 consecutive weeks as maintenance treatment
  * Follow up period: APL-1202 is administered at every 3-month interval if no events occurred in the treatment period and until the occurrence of events or the end of the entire clinical trial Intravesical Epirubicin hydrochloride will be administered once weekly for consecutive 6-8 weeks in the induction period, followed by once monthly in the maintenance period until end of 12 months
  Arms: Placebo

SUMMARY:
To evaluate the clinical efficacy (median event-free survival) of APL-1202 in combination with Epirubicin hydrochloride versus Epirubicin hydrochloride alone in intermediate and high-risk chemo-refractory non-muscle invasive bladder cancer (NMIBC) patients

DETAILED DESCRIPTION:
A multi-center, randomized, double-blind, placebo controlled Phase Ⅲ trial; including 3 stages: screening period, treatment period, and follow-up period.

* Screening period: 6 weeks prior to treatment
* Treatment period:
* Induction period: APL-1202 is administered for 12 consecutive weeks
* Maintenance period: after 12-week drug free period, APL-1202 is administered for another12 consecutive weeks as maintenance treatment
* Follow up period: APL-1202 is administered at every 3-month interval if no events occurred in the treatment period and until the occurrence of events or the end of the entire clinical trial Intravesical Epirubicin hydrochloride will be administered once weekly for consecutive 6-8 weeks in the induction period, followed by once monthly in the maintenance period until end of 12 months

ELIGIBILITY:
Inclusion Criteria:

* Must be informed of the investigational nature of this study and must provide written informed consent
* Age ≥18 years, male or female
* Must have clinically and histologically confirmed recurrent intermediate and high-risk non-muscle invasive transitional cell carcinoma of the bladder after treatment with intravesical chemotherapy. EORTC risk score (according to EUA "NMIBC Guideline" 2015 version) must be ≥ 5: Papilloma alone (or with Cis) or Cis alone No visible tumor after TURBT on tumor lesion
* Medical history of intravesical chemotherapy Subjects who received intravesical chemotherapy prior to enrollment, but didn't receive BCG or other intravesical therapy with immune drugs Subjected who are refractory to the recommended intravesical chemotherapy drugs pirarubicin, epirubicin, doxorubicin, hydroxy camptothecin, mitomycin, or gemcitabine (according to "Guideline of Diagnosis and Treatment of Urological Diseases in China", 2014 version)
* Re-TURBT:

For subjects undergoing secondary TURBT, EORTC risk score must be ≥ 5, which can be assessed based on the results of any TURBTs. The other results will be based on first TURBT For subjects undergoing secondary TURBT, the enrollment time will start from the second TURBT It is recommended to conduct the secondary TURBT under following situations: incomplete first TURBT; no muscle tissue found in the first TURBT specimen, except Ta G1 (low grade) tumor and CIS only; T1 tumor; G3 (high grade) tumor (except CIS) The secondary TURBT is recommended 2-6 weeks, but better at 4 weeks, after the first TURBT

* Willing to provide biopsy specimen for assessment
* ECOG PS ≤ 1, and did not deteriorate in 7 days
* Patients must have normal organ and marrow function within 42 days of study entry (according to normal range in clinical site) Absolute neutrophil count >1.0×109/L Platelets > 100 ×109/L Hemoglobin > 9.0 g/dl Alkaline phosphatase < 2.5 ULN (<10 X ULN in presence of bone metastasis) GFR (Cockcroft-Gault formula calculated) ≥ 50 ml/min INR <1.5, except for subjects receiving warfarin therapy
* Eligibility of patients receiving any medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of APL-1202 will be determined following review of their case by the Principal Investigator
* Female should be either surgically sterilized or menopause or agree to use effective contraceptive measures during treatment
* Male subjects must be surgically sterilized or agreed to use effective contraceptive measures. Subjects must continue to take contraceptive measures within 3 months of the end of the study treatment. The definition of effective contraceptive measures will be based on the Principal Investigator or appointed delegate;
* Expected life expectancy is more than 30 months

Exclusion Criteria:

* TBIL, ALT or AST >1.5 x normal range (according to normal range in clinical sites)
* Urothelial cell carcinoma in upper urethra or ureter
* Received intravesical therapy in last TURBT/cystoscopy prior to enrollment period, but not including immediate intravesical therapy once (the subjects who received the immediate intravesical therapy need to be recorded in e-CRF)
* Received surgery (not includes TURBT/cystoscopy), radiation therapy, or systemic therapy within 6 weeks before enrollment
* Malignancies within 2 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in-situ' of the cervix
* NCI CTCAE grade 3 hemorrhage within 6 weeks of starting study treatment
* Any of the following within 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism
* Hypertension that cannot be controlled by medications
* systolic blood pressure≥140 mmHg and/or diastolic blood pressure≥90mmHg
* Uncontrolled active infections such as acute pneumonia, active hepatitis B, etc.
* Dysphagia or known drug absorption disorders
* Anuria
* One week prior to enrollment, having hematuria
* Active duodenal ulcers, ulcerative colitis and other gastrointestinal diseases or other conditions that the investigator may determine to cause gastrointestinal bleeding or perforation
* Subjects that may increase the risk associated with study participation or study drug administration, judged by investigator, or other severe acute or chronic medical condition or optic nerve disorders may interfere with the interpretation and judgment of study results
* Pregnancy or breastfeeding. Female patients with reproductive potential have a positive pregnancy test prior to enrollment
* Psychological or mental abnormality, subjects are estimated to have insufficient adherence to this clinical study
* Four weeks prior to enrollment, participate in other clinical trials
* Patients who had previously received anthracycline for systemic chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | Up to 30 months
  "Event"is defined as: pathologically confirmed recurrence, progression, or death resulting from bladder cancer

SECONDARY OUTCOMES:
Recurrent-free rate | 24 months
  Recurrent-free rate
Progression-free rate | 24 months
  Progression-free rate
Clinical benefit rate at 12,18, 24 months after enrollment (clinical benefits are defined as the pathological improvement of the recurrence, no high-risk recurrence, progression-free recurrence, no radical therapy and no death) | 24 months
  Clinical benefit rate at 12,18, 24 months after enrollment (clinical benefits are defined as the pathological improvement of the recurrence, no high-risk recurrence, progression-free recurrence, no radical therapy and no death)
Recurrence-free survival | Up to 30 months
  Recurrence-free survival
Progression-free survival | Up to 30 months
  Progression-free survival
Total survival | Up to 30 months
  Total survival

CONTACTS AND LOCATIONS:
Overall Officials: Dingwei Ye, MD,PhD, Principal Investigator — Fudan University; Hanzhong Li, MD,PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No